CLINICAL TRIAL: NCT05815901
Title: A Multi-center, Randomized, Double-blind, Active-controlled, Therapeutic Confirmatory, Phase III Study to Compare and Evaluate the Efficacy and Safety of Epaminurad With Febuxostat in Gout Patients
Brief Title: A Therapeutic Confirmatory Study of Epaminurad Versus Febuxostat in Gout Patients
Acronym: EPIC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JW21301
Record Dates: First submitted 2023-02-27; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Epaminurad 6 mg (Experimental): [Main study period] Epaminurad 6 mg and three matched placebos for 20 weeks. [Extension study period] Epaminurad 6 mg or 9 mg (open label) for 28 weeks.
  Interventions: Drug: Epaminurad 6 mg; Drug: Epaminurad 9 mg placebo; Drug: Febuxostat 40 mg placebo; Drug: Febuxostat 80 mg placebo
- Epaminurad 9 mg (Experimental): [Main study period] Epaminurad 9 mg and three matched placebos for 20 weeks. [Extension study period] Epaminurad 6 mg or 9 mg (open label) for 28 weeks.
  Interventions: Drug: Epaminurad 9 mg; Drug: Epaminurad 6 mg placebo; Drug: Febuxostat 40 mg placebo; Drug: Febuxostat 80 mg placebo
- Febuxostat 40 mg (Active Comparator): [Main study period] Febuxostat 40 mg and three matched placebos for 20 weeks. [Extension study period] Epaminurad 6 mg or 9 mg (open label) for 28 weeks.
  Interventions: Drug: Febuxostat 40 mg; Drug: Epaminurad 6 mg placebo; Drug: Epaminurad 9 mg placebo; Drug: Febuxostat 80 mg placebo
- Febuxostat 80 mg (Active Comparator): [Main study period] Febuxostat 80 mg and three matched placebos for 20 weeks. [Extension study period] Epaminurad 6 mg or 9 mg (open label) for 28 weeks.
  Interventions: Drug: Febuxostat 80 mg; Drug: Epaminurad 6 mg placebo; Drug: Epaminurad 9 mg placebo; Drug: Febuxostat 40 mg placebo

INTERVENTIONS:
Drug: Epaminurad 6 mg — Epaminurad 6 mg tablet
  Arms: Epaminurad 6 mg
Drug: Epaminurad 9 mg — Epaminurad 9 mg tablet
  Arms: Epaminurad 9 mg
Drug: Febuxostat 40 mg — Febuxostat 40 mg tablet
  Arms: Febuxostat 40 mg
Drug: Febuxostat 80 mg — Febuxostat 80 mg tablet
  Arms: Febuxostat 80 mg
Drug: Epaminurad 6 mg placebo — Placebo tablet
  Arms: Epaminurad 9 mg; Febuxostat 40 mg; Febuxostat 80 mg
Drug: Epaminurad 9 mg placebo — Placebo tablet
  Arms: Epaminurad 6 mg; Febuxostat 40 mg; Febuxostat 80 mg
Drug: Febuxostat 40 mg placebo — Placebo tablet
  Arms: Epaminurad 6 mg; Epaminurad 9 mg; Febuxostat 80 mg
Drug: Febuxostat 80 mg placebo — Placebo tablet
  Arms: Epaminurad 6 mg; Epaminurad 9 mg; Febuxostat 40 mg

SUMMARY:
A phase 3 clinical trial to compare and evaluate efficacy and safety of epaminurad with febuxostat in gout patients.

ELIGIBILITY:
Inclusion Criteria:

* for screening

  1. ≥19 to ≤75 years of age at the time of written informed consent
  2. Diagnosed record with gout, or ACR/EULAR 2015 score ≥8
  3. Able and willing to actively participate in TLC programme
  4. Signed ICF for voluntary study participation
* for randomization

  1. sUA level ≥7.0 mg/dL
  2. ACR/EULAR 2015 score ≥8

Exclusion Criteria:

1. Medical history

   Malignant tumor, Urolithiasis within 5 years, Hypersensitivity disease, Lesch-Nyhan syndrome, Hereditary problems, Ischemic heart disease, Prior or planned organ transplant recipient.
2. Concurrent disease or laboratory test abnormality

   Uncontrolled diabetes mellitus, Uncontrolled hypertension, Uncontrolled dyslipidemia, AST or ALT ≥2×ULN, total bilirubin ≥1.5×ULN, eGFR <30 mL/min/1.73m^2, Uncontrolled thyroid dysfunction, HIV, HBV or HCV positive, Drug and alcohol abuse, BMI ≥40 kg/m^2
3. History of gout flare between 2 weeks before written informed consent and immediately before randomization
4. Any cardiovascular abnormalities that might affect the study
5. Prior or planned treatment with xanthine oxidase inhibitors, uricosuric agents, or uricolytic agents
6. Prior or planned treatment with drugs acting on human uric acid transporter 1 or diuretics
7. Prior or planned treatment with intravenous and oral high dose systemic corticosteroids, mercaptopurine, azathioprine, or theophylline
8. Hypersensitivity to the IP (epaminurad or febuxostat)
9. Pregnant or lactating woman.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 588 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with sUA (serum uric acid) <6 mg/dL at the last 3 time points during the main study period | Week 24

SECONDARY OUTCOMES:
Proportion of subjects with sUA <6 mg/dL post-dose at each visit | up to Week 24
Proportion of subjects with sUA <5 mg/dL at the last 3 time points | Week 16, 20, 24
Proportion of subjects with sUA <5 mg/dL post-dose at each visit | up to Week 24
Change from baseline in sUA (mg/dL) at each visit | up to Week 24
Percent change from baseline in sUA at each visit | up to Week 24
Incidence of gout flare post-dose up to Week 24 | up to Week 24
Proportion of subjects who had rescue therapy for gout flare post-dose up to Week 24 | up to Week 24
Adverse events | up to Week 52
  Safety endpoint
Number of subjects with clinical significant results of Laboratory tests | up to Week 52
  Safety endpoint
Number of subjects with clinical significant results of Vital signs | up to Week 52
  Safety endpoint
Number of subjects with clinical significant results of Electrocardiogram | up to Week 52
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, MD, Study Chair — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea